CLINICAL TRIAL: NCT06304844
Title: Assessing the Risk of Chronic Kidney Disease Associated With Metabolic Dysfunction-Associated Fatty Liver Disease in Patients With Type 2 Diabetes Mellitus
Brief Title: Risk of CKD in Diabetic Patients With MAFLD
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Mahmoud Ismail, assistant lecturer - internal medicine department, Sohag University
Other Study IDs: Soh-Med-24-02-06MD
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- diabetic without MAFLD: patients with type 2 DM but has no evidence of MAFLD
- diabetic with MAFLD (high hepatic involvement): patients with type 2 DM and have evidence of MAFLD (according to abdominal ultrasonography) and have high controlled attenuation parameter and liver stiffness measurement in Fibroscan
  Interventions: Diagnostic Test: transient elastography (Fibroscan)
- diabetic with MAFLD (low hepatic involvement): patients with type 2 DM and have evidence of MAFLD (according to abdominal ultrasonography) and have low controlled attenuation parameter and liver stffiness measurement in Fibroscan
  Interventions: Diagnostic Test: transient elastography (Fibroscan)

INTERVENTIONS:
Diagnostic Test: transient elastography (Fibroscan) — conduct fibroscan for patients with (MAFLD by abdominal ultrasonography)
  Groups: diabetic with MAFLD (high hepatic involvement); diabetic with MAFLD (low hepatic involvement)

SUMMARY:
This cross-sectional study of 300 participants investigates the risk of chronic kidney disease (CKD) in individuals with metabolic dysfunction-associated fatty liver disease (MAFLD) and type 2 diabetes. By evaluating hepatic measurements and metabolic markers, the study aims to identify key risk factors for CKD in this population, contributing valuable insights to inform targeted interventions.

DETAILED DESCRIPTION:
investigators plan to enroll 300 participants with type 2 DM to comprehensively investigate the risk of chronic kidney disease (CKD) in individuals diagnosed with metabolic dysfunction-associated fatty liver disease (MAFLD) and type 2 diabetes mellitus.

In this study, the participant population will be grouped based on presence of MAFLD or not into 2 groups, then the group with MAFLD will be subdivided into subgroups based on the degree of hepatic involvement, considering both controlled attenuation parameter (CAP) values for steatosis and liver stiffness measurements for fibrosis via fibro scan device. This grouping strategy aims to categorize individuals into distinct cohorts, such as Low Hepatic Involvement and High Hepatic Involvement groups, facilitating a nuanced exploration of the association between hepatic conditions and the risk of chronic kidney disease (CKD) in the context of metabolic dysfunction-associated fatty liver disease (MAFLD) and type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic patients
* Willing and agreed to be included in the study.

Exclusion Criteria:

* Type 1 diabetic patients or non-diabetic patients.
* Patient with known glomerulonephritis.
* Patient with diagnosis of or clinical features that are suspicious for another systemic disease that commonly causes kidney disease (e.g., connective tissue disorders, HIV).
* Patient with evidence of alternative kidney disease like (Documented obstructive uropathy, etc.)
* Patient with history of kidney transplantation.
* Patient with end stage renal disease or on dialysis.
* Patients with active malignancy.
* Individuals with a history of hepatitis B surface antigen or hepatitis C antibody positivity.
* history of excessive alcohol consumption (⩾30 g/day in men and ⩾20 g/day in women)
* Decompensated liver cirrhosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population for this study comprises individuals diagnosed with type 2 diabetes mellitus either with or without MAFLD. The MAFLD group will encompass individuals meeting standardized diagnostic criteria for MAFLD and having a confirmed diagnosis of type 2 diabetes. Participants with comorbidities, such as viral hepatitis, cirrhosis, and cancers, will be excluded to ensure a focused study population. The chosen sample size of 300 individuals will allow for a robust examination of the prevalence of chronic kidney disease and associated risk factors within this specific cohort.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-04-20 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Determine the number of participant with eGFR<60 ml/min/1.73 m2 or albuminuria (urinary albumin-to-creatinine ratio (ACR) ⩾3 mg/mmol) in patients with type 2 DM and MAFLD | 6 months from the start of participants recruitment
  utilizing standardized diagnostic criteria for CKD including estimated glomerular filtration rate (eGFR) and urinary albumin-to-creatinine ratio (UACR)

IPD SHARING:
Plan to Share IPD: No